CLINICAL TRIAL: NCT06666972
Title: Evaluation of Different Diagnostic Methods of Tuberculosis in Assiut University Hospital
Brief Title: Evaluation of Different Diagnostic Methods of Tuberculosis in Assiut University Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdou Mahmoud, clinical pathology specialist, Assiut University
Other Study IDs: TB diagnosis in AssiutU
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Tuberculosis Diagnosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PCR MTB/NTM — • The Polymerase chain reaction (PCR) MTB/NTM MDR-TB test is an innovative technology that offers a cutting-edge approach to the precise diagnosis of tuberculosis and nontuberculous mycobacterial infections (NTM).

SUMMARY:
* Detection of sensitivity and specificity of microscopic examination and Molecular studies using polymerase chain reaction (PCR) Mycobacterium tuberculosis (MTB)/ non tuberculous mycobacterium (NTM) MDR-TB compared to culture which is the gold standard technique in the diagnosis of TB to reach the most reliable one for better health care service.
* Assess the prevalence of tuberculosis cases among clinically suspected cases admitted to the hospital throughout the selected study period.

DETAILED DESCRIPTION:
Tuberculosis (TB) is an infectious disease of global public health importance caused by the M. tuberculosis complex. Alarmingly, the disease has worsened with the emergence of multidrug-resistant strains of tuberculosis (MDR-TB).

Annually, it is estimated that approximately 450,000 new cases of MDR-TB occur according to a report from 2021.

There is an alarming increase in the global incidence rate of tuberculosis in the year 2021 after covid-19 pandemic, reversing the downward trend maintained in previous decades. In parallel, there is a rise in cases of drug-resistant tuberculosis.

Early diagnosis and appropriate treatment of tuberculosis are essential public health priorities. In this context, microbiology laboratories play a vital role in the rapid and accurate detection of tuberculosis and drug resistance.

Accurate and prompt diagnosis of TB is essential for the control and management of the disease, but there are numerous factors that affect the effectiveness of this process. These problems include the difficulty of correctly diagnosing latent and active forms of TB, the lack of precise protocols for different types of TB, and the difficulty of accessing diagnostic facilities in regions with limited resources.

Laboratory diagnosis of pulmonary tuberculosis is essential in combating the disease, with a significant role in patient management and isolation of contagious cases. In many developing countries with a high incidence of TB, advanced diagnostic methods and drug susceptibility testing are rarely available.

Given its substantial influence on global health, it is imperative that the investigators continue researching and developing innovative techniques and technologies to better the detection and treatment of tuberculosis.

In our study, the investigators try to compare between different available tests to diagnose TB for better treatment and health care service.

ELIGIBILITY:
Inclusion Criteria:

* Patients with signs and symptoms of tuberculosis (suspected cases)
* Patients diagnosed with tuberculosis.

Exclusion Criteria:

* Patients with pulmonary infections other than TB

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with signs and symptoms of tuberculosis (suspected cases) and Patients diagnosed with tuberculosis of both sexes admitted to Assiut university hospitals
Sampling Method: Non-Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
*Compare between different available tests to reach the most reliable one for better health care service. | two years
  *Detection of sensitivity and specificity of microscopic examination and Molecular studies using PCR MTB/NTM MDR-TB compared to culture which is the gold standard technique in the diagnosis of TB to reach the most reliable one for better health care service.

SECONDARY OUTCOMES:
*Assess the prevalence of tuberculosis cases among clinically suspected cases admitted to the hospital throughout the selected study period. | two years

REFERENCES:
- [Background] Rakotosamimanana N, Rabodoarivelo MS, Palomino JC, Martin A, Razanamparany VR. Exploring tuberculosis by molecular tests on DNA isolated from smear microscopy slides. Int J Infect Dis. 2017 Mar;56:248-252. doi: 10.1016/j.ijid.2016.12.005. Epub 2016 Dec 12. PMID 27979786